CLINICAL TRIAL: NCT02054130
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of MEDI9929 in Adult Subjects With Inadequately Controlled, Severe Asthma
Brief Title: Study to Evaluate the Efficacy and Safety of MEDI9929 (AMG 157) in Adult Subjects With Inadequately Controlled, Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-RI-MEDI9929-1146; 2013-003269-33 (EudraCT Number)
Record Dates: First submitted 2013-12-04; First posted 2014-02-04 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo matched to MEDI9929 subcutaneously once every 2 weeks from Day 1 to Week 50.
  Interventions: Drug: Placebo
- MEDI9929 70 mg (Experimental): Participants received 70 milligram (mg) of MEDI9929 subcutaneously once every 4 weeks from Day 1 to Week 48 along with subcutaneous placebo once every 4 weeks from Week 2 to Week 50.
  Interventions: Drug: MEDI9929 70 mg
- MEDI9929 210 mg (Experimental): Participants received 210 mg of MEDI9929 subcutaneously once every 4 weeks from Day 1 to Week 48 along with subcutaneous placebo once every 4 weeks from Week 2 to Week 50.
  Interventions: Drug: MEDI9929 210 mg
- MEDI9929 280 mg (Experimental): Participants received 280 mg of MEDI9929 subcutaneously once every 2 weeks from Day 1 to Week 50.
  Interventions: Drug: MEDI9929 280 mg

INTERVENTIONS:
Drug: Placebo — Participants received placebo matched to MEDI9929 subcutaneously once every 2 weeks from Day 1 to Week 50.
  Arms: Placebo
Drug: MEDI9929 70 mg — Participants received 70 milligram (mg) of MEDI9929 subcutaneously once every 4 weeks from Day 1 to Week 48 along with subcutaneous placebo once every 4 weeks from Week 2 to Week 50.
  Arms: MEDI9929 70 mg
Drug: MEDI9929 210 mg — Participants received 210 mg of MEDI9929 subcutaneously once every 4 weeks from Day 1 to Week 48 along with subcutaneous placebo once every 4 weeks from Week 2 to Week 50.
  Arms: MEDI9929 210 mg
Drug: MEDI9929 280 mg — Participants received 280 mg of MEDI9929 subcutaneously once every 2 weeks from Day 1 to Week 50.
  Arms: MEDI9929 280 mg

SUMMARY:
The primary objective of the study is to evaluate the effect of 3 dose levels of MEDI9929 (AMG 157) on asthma exacerbations in adult subjects with inadequately controlled, severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 75
* Body mass index (BMI) between 18-40 kg/m2 and weight greater than or equal 40 kg
* Documented physician-diagnosed asthma - Subjects must have received a physician-prescribed asthma controller regimen with medium- or high-dose inhaled corticosteroids (ICS) plus long acting β2 agonist (LABA) -If on asthma controller medications in addition to ICS plus LABA, the dose of the other asthma controller medications (leukotriene receptor inhibitors, theophylline, secondary ICS, long-acting anti-muscarinics (LAMA), cromones, or maintenance oral prednisone or equivalent up to a maximum of 10 mg daily or 20 mg every other day for the maintenance treatment of asthma) must be stable. -Subjects must have a documented history of at least 2 asthma exacerbation events OR at least 1 severe asthma exacerbation resulting in hospitalization within the 12 months prior to first study visit.

Exclusion Criteria:

* Diagnosis of vocal cord dysfunction, reactive airways dysfunction syndrome, hyperventilation and panic attacks, or other mimics of asthma.
* Current smokers or subjects with a smoking history of ≥ 10 pack years
* Former smokers with < 10 pack years must have stopped for at least 1 year to be eligible.
* Any concomitant respiratory disease that in the opinion of the investigator and/or medical monitor will interfere with the evaluation of the investigational product or interpretation of subject safety or study results (eg, chronic obstructive pulmonary disease, cystic fibrosis, pulmonary fibrosis, bronchiectasis, allergic bronchopulmonary aspergillosis, Churg-Strauss syndrome).
* Evidence of active liver disease.
* History of Cancer, except for basal cell carcinoma or insitu carcinoma of the cervix treated with apparent success with curative therapy or other malignancies are eligible provided that curative therapy was completed -Known history of active tuberculosis (TB)
* History of anaphylaxis to any biologic therapy
* Positive medical history for hepatitis B or C
* Subject with human immunodeficiency virus (HIV) or subject taking antiretroviral medications, as determined by medical history and/or subject's verbal report.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (86):
- United States (15):
  - Research Site, Los Angeles, California
  - Research Site, Miami, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Dublin, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Velingrad
- Czechia (5):
  - Research Site, Brandýs nad Labem
  - Research Site, Hradec Králové
  - Research Site, Mladá Boleslav
  - Research Site, Prague
  - Research Site, Strakonice
- Hungary (12):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Csorna
  - Research Site, Debrecen
  - Research Site, Farkasgyepü
  - Research Site, Gödöllő
  - Research Site, Komárom
  - Research Site, Mátészalka
  - Research Site, Nagykanizsa
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Törökbálint
- Israel (7):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Litwinsky
- Japan (12):
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Kiyose-shi
  - Research Site, Kurume-shi
  - Research Site, Maebashi
  - Research Site, Ora-gun
  - Research Site, Sagamihara-shi
  - Research Site, Saitama-Ken
  - Research Site, Sapporo
  - Research Site, Taito-ku
  - Research Site, Toshima-ku
  - Research Site, Yokkaichi-shi
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Rēzekne
  - Research Site, Riga
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Klaipėda
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
- Slovakia (12):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Ilava
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Spišská Nová Ves
  - Research Site, Štúrovo
  - Research Site, Šurany
  - Research Site, Topoľčany
  - Research Site, Zvolen
- South Africa (3):
  - Research Site, Durban
  - Research Site, Middelburg
  - Research Site, Pretoria
- Ukraine (9):
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Mykolayiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Suprunivka Vil., Poltava Regio
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya

REFERENCES:
- [Background] Corren J, Parnes JR, Wang L, Mo M, Roseti SL, Griffiths JM, van der Merwe R. Tezepelumab in Adults with Uncontrolled Asthma. N Engl J Med. 2017 Sep 7;377(10):936-946. doi: 10.1056/NEJMoa1704064. PMID 28877011
- [Derived] Feleszko W, Caminati M, Gern JE, Johnston SL, Marchese C, Clarke D, Ambrose CS, Lindsley AW. Effect of tezepelumab on asthma exacerbations co-occurring with infection-attributed acute respiratory illnesses. Ann Allergy Asthma Immunol. 2026 Jan;136(1):61-65.e1. doi: 10.1016/j.anai.2025.09.015. Epub 2025 Oct 8. PMID 41072729
- [Derived] Pavord ID, Brightling CE, Korn S, Martin NL, Ponnarambil SS, Molfino NA, Parnes JR, Ambrose CS. Tezepelumab can Restore Normal Lung Function in Patients with Severe, Uncontrolled Asthma: Pooled Results from the PATHWAY and NAVIGATOR Studies. Pulm Ther. 2025 Jun;11(2):315-325. doi: 10.1007/s41030-025-00294-2. Epub 2025 Apr 26. PMID 40285963
- [Derived] Corren J, Menzies-Gow A, Bimmel J, McGuinness A, Almqvist G, Bowen K, Griffiths JM, Ponnarambil S, Bourdin A, Israel E, Colice G, Brightling CE, Wechsler ME; PATHWAY and NAVIGATOR study investigators. Tezepelumab for the treatment of severe asthma: a plain language summary of the PATHWAY and NAVIGATOR studies. Immunotherapy. 2023 Nov;15(16):1327-1340. doi: 10.2217/imt-2023-0109. Epub 2023 Sep 29. PMID 37772607
- [Derived] Corren J, Menzies-Gow A, Chupp G, Israel E, Korn S, Cook B, Ambrose CS, Hellqvist A, Roseti SL, Molfino NA, Llanos JP, Martin N, Bowen K, Griffiths JM, Parnes JR, Colice G. Efficacy of Tezepelumab in Severe, Uncontrolled Asthma: Pooled Analysis of the PATHWAY and NAVIGATOR Clinical Trials. Am J Respir Crit Care Med. 2023 Jul 1;208(1):13-24. doi: 10.1164/rccm.202210-2005OC. PMID 37015033
- [Derived] Corren J, Pham TH, Garcia Gil E, Salapa K, Ren P, Parnes JR, Colice G, Griffiths JM. Baseline type 2 biomarker levels and response to tezepelumab in severe asthma. Allergy. 2022 Jun;77(6):1786-1796. doi: 10.1111/all.15197. Epub 2022 Feb 9. PMID 34913186
- [Derived] Corren J, Ambrose CS, Salapa K, Roseti SL, Griffiths JM, Parnes JR, Colice G. Efficacy of Tezepelumab in Patients with Severe, Uncontrolled Asthma and Perennial Allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4334-4342.e6. doi: 10.1016/j.jaip.2021.07.045. Epub 2021 Aug 3. PMID 34358701
- [Derived] Ly N, Zheng Y, Griffiths JM, van der Merwe R, Agoram B, Parnes JR, Roskos L. Pharmacokinetic and Pharmacodynamic Modeling of Tezepelumab to Guide Phase 3 Dose Selection for Patients With Severe Asthma. J Clin Pharmacol. 2021 Jul;61(7):901-912. doi: 10.1002/jcph.1803. Epub 2021 Jan 16. PMID 33368307
- [Derived] Corren J, Garcia Gil E, Griffiths JM, Parnes JR, van der Merwe R, Salapa K, O'Quinn S. Tezepelumab improves patient-reported outcomes in patients with severe, uncontrolled asthma in PATHWAY. Ann Allergy Asthma Immunol. 2021 Feb;126(2):187-193. doi: 10.1016/j.anai.2020.10.008. Epub 2020 Oct 23. PMID 33169672
- See also: CD-RI-MEDI9929-1146_Protocol_Synopsis_Amendment_3_Redacted_04.03.17 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1887&filename=CD-RI-MEDI9929-1146_Protocol_Synopsis_Amendment_3_Redacted_04.03.17.pdf
- See also: CD-RI-MEDI9929-1146_Protocol_Synopsis_Redacted_06.23.17 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1887&filename=CD-RI-MEDI9929-1146_Protocol_Synopsis_Redacted_06.23.17.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 19Dec2013 to 01Mar2017 across 12 countries (United States, Slovakia, Bulgaria, Czech Republic, Hungary, Israel, Japan, Latvia, Lithuania, Serbia, South Africa, and Ukraine). A total of 918 participants were recruited in the study.
Pre-assignment Details: Of 918 participants, 334 were considered screen failures and 584 participants were randomized. Of which, all populations excluded 34 participants from one site due to non-compliance of the principles of Good Clinical Practice.
Period: Overall Study
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Started | 138 | 138 | 137 | 137
Completed | 130 | 127 | 122 | 115
Not Completed | 8 | 11 | 15 | 22
Not completed — Withdrawal by Subject | 4 | 4 | 7 | 10
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Missed dose | 4 | 6 | 7 | 10

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population included participants who are randomized and received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg | Total
Number analyzed (Participants) | 138 | 138 | 137 | 137 | 550
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.32 (11.71) | 50.80 (12.36) | 52.66 (12.67) | 50.43 (12.25) | 51.55 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 89 | 87 | 91 | 361
  Male | 44 | 49 | 50 | 46 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 137 | 138 | 136 | 135 | 546
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 3 | 5 | 5 | 19
  Black or African American | 6 | 4 | 3 | 6 | 19
  White | 123 | 131 | 128 | 122 | 504
  Other | 2 | 0 | 0 | 2 | 4
  Multiple Categories Checked | 1 | 0 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Annualized Asthma Exacerbation Rate (AER) Through Week 52
Description: Asthma exacerbation is defined as worsening of asthma that leads to any of the following: use of systemic corticosteroids for at least 3 days, an emergency department visit due to asthma that required systemic corticosteroids, and an inpatient hospitalization due to asthma. The annual AER was presented as the total number of exacerbations for the treatment group divided by the total duration of person follow-up.
Time Frame: Week 0 (Day 1) up to Week 52
Population: Intent-to-treat population included all participants who are randomized and received any study drug.
Measure: Number (95% Confidence Interval); unit: events per person-year
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
events per person-year | 0.72 [0.59 to 0.88] | 0.27 [0.19 to 0.38] | 0.20 [0.13 to 0.30] | 0.23 [0.16 to 0.34]
Statistical Analysis 1: Comparison: Placebo vs MEDI9929 70 mg; Test type: Superiority; p < 0.001, Negative binomial regression; Rate ratio = 0.38, 95% CI 2-sided [0.23 to 0.63]
Statistical Analysis 2: Comparison: Placebo vs MEDI9929 210 mg; Test type: Superiority; p < 0.001, Negative binomial regression; Rate ratio = 0.29, 95% CI 2-sided [0.16 to 0.51]
Statistical Analysis 3: Comparison: Placebo vs MEDI9929 280 mg; Test type: Superiority; p < 0.001, Negative bnomial regression; Rate ratio = 0.34, 95% CI 2-sided [0.20 to 0.58]

2. Secondary Outcome: Reduction in AER on Subpopulations at Week 52
Description: Asthma exacerbation is defined as worsening of asthma that leads to any of the following: use of systemic corticosteroids for at least 3 days, an emergency department visit due to asthma that required systemic corticosteroids, and an inpatient hospitalization due to asthma. Reduction in AER was evaluated in pre-specified subpopulations (blood eosinophil count [eosinophilic and non-eosinophilic], T helper cell 2 [Th2] status [high and low], Fraction of exhaled nitric oxide [FENO] [high and low], serum periostin [high and low], current post bronchodilator forced expiratory volume in 1 second [Post-BD FEV1] reversibility- yes, allergic and non-allergic) of asthma. The annual AER was presented as the total number of exacerbations for the treatment group divided by the total duration of person follow-up. Also, the high or low was determined using median value.
Time Frame: Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: events per person-year
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
events per person-year
  Blood Eosinophil Count -Eosinophilic: number analyzed (Participants) | 78 | 80 | 76 | 76
  Blood Eosinophil Count -Eosinophilic | 0.78 [0.59 to 1.00] | 0.29 [0.18 to 0.43] | 0.26 [0.16 to 0.42] | 0.21 [0.12 to 0.35]
  Blood Eosinophil Count -Non-Eosinophilic: number analyzed (Participants) | 60 | 58 | 61 | 61
  Blood Eosinophil Count -Non-Eosinophilic | 0.65 [0.46 to 0.89] | 0.25 [0.14 to 0.42] | 0.14 [0.06 to 0.27] | 0.26 [0.14 to 0.43]
  Th2 Status - High: number analyzed (Participants) | 75 | 62 | 65 | 62
  Th2 Status - High | 0.62 [0.45 to 0.83] | 0.33 [0.20 to 0.50] | 0.25 [0.14 to 0.41] | 0.21 [0.11 to 0.36]
  Th2 Status - Low: number analyzed (Participants) | 62 | 75 | 70 | 74
  Th2 Status - Low | 0.86 [0.64 to 1.13] | 0.23 [0.14 to 0.37] | 0.15 [0.07 to 0.28] | 0.26 [0.15 to 0.41]
  FENO - High: number analyzed (Participants) | 70 | 72 | 68 | 64
  FENO - High | 0.94 [0.72 to 1.20] | 0.32 [0.20 to 0.48] | 0.20 [0.11 to 0.35] | 0.20 [0.10 to 0.35]
  FENO - Low: number analyzed (Participants) | 67 | 65 | 67 | 69
  FENO - Low | 0.51 [0.36 to 0.72] | 0.23 [0.13 to 0.38] | 0.21 [0.11 to 0.36] | 0.28 [0.16 to 0.44]
  Serum Periostin - High: number analyzed (Participants) | 69 | 63 | 73 | 68
  Serum Periostin - High | 0.78 [0.59 to 1.02] | 0.29 [0.17 to 0.45] | 0.19 [0.10 to 0.33] | 0.19 [0.10 to 0.32]
  Serum Periostin - Low: number analyzed (Participants) | 69 | 74 | 63 | 66
  Serum Periostin - Low | 0.66 [0.48 to 0.89] | 0.27 [0.16 to 0.42] | 0.22 [0.12 to 0.38] | 0.30 [0.18 to 0.47]
  Current Post-BD FEV1 Reversibility-Yes: number analyzed (Participants) | 126 | 123 | 114 | 125
  Current Post-BD FEV1 Reversibility-Yes | 0.60 [0.47 to 0.75] | 0.26 [0.18 to 0.37] | 0.17 [0.10 to 0.27] | 0.21 [0.14 to 0.32]
  Allergic: number analyzed (Participants) | 80 | 68 | 77 | 71
  Allergic | 0.75 [0.57 to 0.97] | 0.25 [0.15 to 0.40] | 0.14 [0.07 to 0.26] | 0.23 [0.13 to 0.38]
  Non-Allergic: number analyzed (Participants) | 50 | 60 | 50 | 58
  Non-Allergic | 0.65 [0.44 to 0.91] | 0.23 [0.12 to 0.39] | 0.26 [0.13 to 0.45] | 0.22 [0.11 to 0.38]

3. Secondary Outcome: Change From Baseline in Pre-bronchodilator (Pre-BD) Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) at Week 52
Description: Forced expiratory volume in 1 second and forced vital capacity measures taken before bronchodilator use were reported.
Time Frame: Baseline (Week 0 [Day 1]) to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Liter
  Change from Baseline in Pre-BD FEV1: number analyzed (Participants) | 131 | 130 | 121 | 116
  Change from Baseline in Pre-BD FEV1 | 0.071 (0.405) | 0.200 (0.432) | 0.210 (0.433) | 0.245 (0.411)
  Change from Baseline in Pre-BD FVC: number analyzed (Participants) | 131 | 130 | 121 | 116
  Change from Baseline in Pre-BD FVC | 0.068 (0.477) | 0.244 (0.560) | 0.202 (0.616) | 0.197 (0.484)

4. Secondary Outcome: Change From Baseline in FEV1 on Subpopulations at Week 52
Description: Forced expiratory volume in one second (FEV1) was evaluated in pre-specified subpopulations of asthma. The data presented in the below table for this outcome measure is for pre-bronchodilator FEV1.
Time Frame: Baseline and up to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Liters
  Blood Eosinophil Count -Eosinophilic: number analyzed (Participants) | 76 | 77 | 66 | 63
  Blood Eosinophil Count -Eosinophilic | -0.045 (0.080) | 0.118 (0.083) | 0.125 (0.086) | 0.160 (0.080)
  Blood Eosinophil Count -Non-Eosinophilic: number analyzed (Participants) | 55 | 53 | 55 | 53
  Blood Eosinophil Count -Non-Eosinophilic | -0.072 (0.105) | -0.030 (0.112) | 0.008 (0.106) | 0.011 (0.108)
  Th2 Status - High: number analyzed (Participants) | 73 | 59 | 57 | 53
  Th2 Status - High | -0.058 (0.101) | 0.037 (0.109) | 0.052 (0.107) | 0.182 (0.104)
  Th2 Status - Low: number analyzed (Participants) | 57 | 70 | 62 | 62
  Th2 Status - Low | -0.052 (0.085) | 0.103 (0.086) | 0.103 (0.088) | 0.062 (0.086)
  FENO - High: number analyzed (Participants) | 65 | 66 | 60 | 54
  FENO - High | -0.054 (0.078) | 0.093 (0.084) | 0.137 (0.083) | 0.155 (0.079)
  FENO - Low: number analyzed (Participants) | 65 | 63 | 59 | 59
  FENO - Low | 0.027 (0.074) | 0.115 (0.076) | 0.095 (0.073) | 0.133 (0.075)
  Serum Periostin - High: number analyzed (Participants) | 67 | 61 | 65 | 61
  Serum Periostin - High | -0.017 (0.088) | 0.147 (0.094) | 0.207 (0.092) | 0.185 (0.089)
  Serum Periostin - Low: number analyzed (Participants) | 64 | 68 | 55 | 52
  Serum Periostin - Low | -0.040 (0.090) | 0.060 (0.093) | -0.013 (0.093) | 0.064 (0.089)
  Current Post-BD FEV1 Reversibility - Yes: number analyzed (Participants) | 120 | 117 | 102 | 105
  Current Post-BD FEV1 Reversibility - Yes | -0.081 (0.075) | 0.052 (0.077) | 0.049 (0.077) | 0.066 (0.073)
  Allergic: number analyzed (Participants) | 75 | 65 | 70 | 57
  Allergic | -0.047 (0.073) | 0.131 (0.081) | 0.084 (0.077) | 0.065 (0.076)
  Non-Allergic: number analyzed (Participants) | 48 | 56 | 42 | 52
  Non-Allergic | -0.037 (0.131) | 0.050 (0.123) | 0.148 (0.129) | 0.164 (0.123)

5. Secondary Outcome: Change From Baseline in Post-bronchodilator (Post-BD) FEV1 and FVC at Week 52
Description: Forced expiratory volume in 1 second and forced vital capacity measures taken after bronchodilator use were reported.
Time Frame: Baseline (Week 0 [Day 1]) to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Liter
  Change from Baseline in Post-BD FEV1: number analyzed (Participants) | 130 | 130 | 121 | 115
  Change from Baseline in Post-BD FEV1 | -0.064 (0.352) | 0.117 (0.389) | 0.099 (0.449) | 0.128 (0.415)
  Change from Baseline in Post-BD FVC: number analyzed (Participants) | 130 | 130 | 121 | 115
  Change from Baseline in Post-BD FVC | -0.092 (0.353) | 0.088 (0.439) | 0.092 (0.515) | 0.083 (0.435)

6. Secondary Outcome: Change From Baseline in Overall Symptoms Score on Subpopulations at Week 52
Description: Asthma symptoms during night time and daytime are recorded by the participant in the asthma daily diary. Overall symptom score is the average of scores of daytime severity, daytime frequency, and nighttime severity symptoms. The daytime frequency and severity items are scored from 0 to 4, where a higher score indicates greater frequency/severity and nighttime severity item is scored from 0 to 4 , where a higher score indicates greater severity. Overall symptom score ranges from 0 to 4, where lower score indicates better asthma symptom while, higher score indicates worse asthma symptom.
Time Frame: Baseline and up to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Units on a scale
  Blood Eosinophil Count -Eosinophilic: number analyzed (Participants) | 70 | 72 | 58 | 54
  Blood Eosinophil Count -Eosinophilic | -0.57 (0.07) | -0.62 (0.07) | -0.78 (0.07) | -0.72 (0.07)
  Blood Eosinophil Count -Non-Eosinophilic: number analyzed (Participants) | 48 | 47 | 47 | 49
  Blood Eosinophil Count -Non-Eosinophilic | -0.49 (0.08) | -0.60 (0.08) | -0.56 (0.08) | -0.72 (0.08)
  Th2 Status - High: number analyzed (Participants) | 65 | 54 | 51 | 48
  Th2 Status - High | -0.54 (0.07) | -0.65 (0.08) | -0.62 (0.08) | -0.75 (0.08)
  Th2 Status - Low: number analyzed (Participants) | 52 | 64 | 52 | 54
  Th2 Status - Low | -0.50 (0.08) | -0.57 (0.07) | -0.72 (0.08) | -0.71 (0.08)
  FENO - High: number analyzed (Participants) | 59 | 60 | 49 | 44
  FENO - High | -0.52 (0.08) | -0.68 (0.07) | -0.75 (0.08) | -0.72 (0.08)
  FENO - Low: number analyzed (Participants) | 59 | 58 | 54 | 56
  FENO - Low | -0.54 (0.07) | -0.55 (0.07) | -0.59 (0.08) | -0.71 (0.07)
  Serum Periostin - High: number analyzed (Participants) | 63 | 57 | 56 | 54
  Serum Periostin - High | -0.48 (0.07) | -0.54 (0.08) | -0.84 (0.08) | -0.74 (0.08)
  Serum Periostin - Low: number analyzed (Participants) | 55 | 61 | 48 | 46
  Serum Periostin - Low | -0.58 (0.07) | -0.63 (0.07) | -0.47 (0.08) | -0.69 (0.07)
  Current Post-BD FEV1 Reversibility - Yes: number analyzed (Participants) | 108 | 106 | 87 | 92
  Current Post-BD FEV1 Reversibility - Yes | -0.55 (0.05) | -0.60 (0.06) | -0.64 (0.06) | -0.71 (0.06)
  Allergic: number analyzed (Participants) | 66 | 56 | 60 | 48
  Allergic | -0.53 (0.07) | -0.59 (0.07) | -0.63 (0.07) | -0.67 (0.07)
  Non-Allergic: number analyzed (Participants) | 46 | 55 | 36 | 47
  Non-Allergic | -0.50 (0.09) | -0.60 (0.08) | -0.72 (0.09) | -0.85 (0.08)

7. Secondary Outcome: Change From Baseline in Asthma Symptoms Measured by Asthma Daily Diary at Week 52
Description: Asthma symptoms during night time and daytime are recorded by the participant in the asthma daily diary. Symptom score values for night time assessment is 0 (no asthma symptom) to 3 (unable to sleep because of asthma) and symptom score values for day time assessment is 0 (no asthma symptom) to 3 (unable to do normal activities due to asthma). Total asthma symptom score is the sum of the daytime and night time score (0 to 6). Lower score (0) is indicating better asthma symptom, while higher score (6) is indicating worse asthma symptom.
Time Frame: Baseline (Week 0 [Day 1]) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Units on a scale
  Daytime Severity: number analyzed (Participants) | 118 | 119 | 105 | 103
  Daytime Severity | -0.483 (0.700) | -0.657 (0.726) | -0.669 (0.640) | -0.680 (0.688)
  Daytime Frequency: number analyzed (Participants) | 118 | 119 | 105 | 103
  Daytime Frequency | -0.493 (0.792) | -0.598 (0.837) | -0.727 (0.753) | -0.754 (0.752)
  Nighttime Severity: number analyzed (Participants) | 118 | 119 | 105 | 103
  Nighttime Severity | -0.643 (0.799) | -0.616 (0.687) | -0.807 (0.699) | -0.662 (0.730)

8. Secondary Outcome: Change From Baseline in Asthma Symptoms Measured by Asthma Control Questionnaire (ACQ-6) Score at Week 52
Description: The ACQ is a patient-reported questionnaire assessing asthma symptoms (ie, night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use and FEV1. The ACQ-6 is a shortened version of the ACQ that omits the FEV1 measurement from the original ACQ score. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled).
Time Frame: Baseline (Week 0 [Day 1]) and Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Units on a scale | -0.89 (0.91) | -1.24 (0.94) | -1.17 (1.00) | -1.19 (1.00)

9. Secondary Outcome: Rate of Severe Asthma Exacerbation Through Week 52
Description: A severe asthma exacerbation is defined as an event that resulted in hospitalization. The severe AER was presented as the total number of exacerbations for the treatment group divided by the total duration of person follow-up.
Time Frame: Week 0 (Day 1) up to Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Number (95% Confidence Interval); unit: events per person-year
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
events per person-year | 0.14 [0.08 to 0.22] | 0.04 [0.01 to 0.09] | 0.02 [0.00 to 0.07] | 0.03 [0.01 to 0.08]

10. Secondary Outcome: Time to First Asthma Exacerbation Through Week 52
Description: Asthma exacerbation is defined as worsening of asthma that leads to use of systemic corticosteroids for at least 3 days, an emergency department visit due to asthma that required systemic corticosteroids, and an inpatient hospitalization due to asthma. Time to first asthma exacerbation was reported.
Time Frame: Week 0 (Day 1) through Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Days | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations. | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations. | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations. | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations.

11. Secondary Outcome: Time to First Severe Asthma Exacerbation Through Week 52
Description: Asthma exacerbation is defined as worsening of asthma that leads to use of systemic corticosteroids for at least 3 days, an emergency department visit due to asthma that required systemic corticosteroids, and an inpatient hospitalization due to asthma. Time to first severe asthma exacerbations (hospitalization) were reported.
Time Frame: Week 0 (Day 1) through Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Days | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations. | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations. | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations. | NA [NA to NA] — Median survival time was not estimable as less than 50% participants had exacerbations.

12. Secondary Outcome: Number of Participants With at Least One Asthma Exacerbations Through Week 52
Description: Asthma exacerbation is defined as worsening of asthma that leads to use of systemic corticosteroids for at least 3 days, an emergency department visit due to asthma that required systemic corticosteroids, and an inpatient hospitalization due to asthma.
Time Frame: Week 0 (Day 1) through Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants | 43 | 30 | 21 | 25

13. Secondary Outcome: Number of Participants With at Least One Severe Asthma Exacerbations Through Week 52
Description: Asthma exacerbation is defined as worsening of asthma that leads to use of systemic corticosteroids for at least 3 days, an emergency department visit due to asthma that required systemic corticosteroids, and an inpatient hospitalization due to asthma. Participants with severe asthma exacerbations (hospitalization) were reported.
Time Frame: Week 0 (Day 1) through Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants | 9 | 5 | 3 | 4

14. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ [S]) Overall Score at Week 52
Description: The AQLQ(S) +12 is a 32-item questionnaire that measures the health-related quality of life experienced by asthma participants. The questionnaire comprises 4 separate domains (symptoms, activity limitations, emotional function, and environmental stimuli) scaled on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment).
Time Frame: Baseline (Week 0 [Day 1]) and Week 52
Population: Intent-to-treat population included participants who are randomized and received any study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Units on a scale | 1.04 (1.11) | 1.19 (0.90) | 0.93 (1.03) | 1.13 (1.13)

15. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions 5 Level Version (EQ-5D-5L) Health State Evaluation at Week 52
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. The first component is a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1. A higher score indicates better health state. The second component is a self-perceived health score which is assessed using a visual analogue scale (VAS) that ranged from 0 to 100, where 0 indicated the worst health you can imagine and 100 indicated the best health you can imagine.
Time Frame: Baseline (Week 0 [Day 1]) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Units on a scale
  Health State Valuation: number analyzed (Participants) | 38 | 41 | 33 | 40
  Health State Valuation | 0.1051 (0.1511) | 0.0752 (0.2179) | 0.0729 (0.1624) | 0.0395 (0.1935)
  Visual Analog Scale | 13.8 (17.6) | 14.0 (16.4) | 12.0 (18.0) | 12.3 (18.0)

16. Secondary Outcome: Total Amount of Study Drug Exposure
Description: The total amount of study drug exposure (in milligram) for the entire study period was summarized.
Time Frame: Week 0 (Day 1) through Week 52
Population: As-treated population included all participants who received any study drug.
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 137 | 137
Milligram | 877.0 (116.9) | 2493.9 (640.4) | 6574.9 (1630.2)

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event is any unfavourable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with use of medicinal product, whether or not considered related to medicinal product. Serious adverse event is any adverse event that resulted in death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug, for the period until and including the follow-up period (Week 64).
Time Frame: Day 1 upto Week 64
Population: As-treated population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants
  TEAEs | 91 | 93 | 90 | 89
  TESAEs | 18 | 17 | 13 | 18

18. Secondary Outcome: Number of Participants With TEAEs Related to Vital Sign Parameters
Description: Adverse events observed in participants with clinically significant vital signs abnormalities were assessed.
Time Frame: Day 1 upto Week 64
Population: As-treated population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants
  Blood pressure diastolic increased | 0 | 1 | 0 | 0
  Blood pressure increased | 1 | 2 | 1 | 0
  Heart rate increased | 0 | 0 | 0 | 1
  Hypertension | 7 | 7 | 5 | 6
  Hypertensive crisis | 0 | 0 | 0 | 1
  Hypotension | 0 | 0 | 0 | 2
  Pyrexia | 0 | 2 | 2 | 0
  Respiratory rate increased | 0 | 0 | 0 | 1

19. Secondary Outcome: Number of Participants With TEAEs Related to Clinical Laboratory Evaluation
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Laboratory evaluations of blood and urine samples were performed.
Time Frame: Day 1 upto Week 64
Population: As-treated population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants
  Anaemia | 0 | 0 | 0 | 1
  Leukopenia | 0 | 1 | 0 | 0
  Lymphopenia | 0 | 1 | 0 | 0
  Neutropenia | 0 | 1 | 0 | 0
  Thrombocytopenia | 0 | 1 | 0 | 0
  Dyslipidaemia | 0 | 1 | 0 | 0
  Hepatic enzyme increased | 0 | 0 | 1 | 0
  Hypercholesterolaemia | 0 | 0 | 1 | 0
  Hyperuricaemia | 0 | 0 | 1 | 0
  Hypokalaemia | 0 | 0 | 1 | 0
  Vitamin D deficiency | 0 | 0 | 1 | 0
  Hematuria | 1 | 0 | 1 | 0

20. Secondary Outcome: Number of Participants With TEAEs Related to Electrocardiogram Evaluations
Description: Adverse events observed in participants with clinically significant electrocardiogram abnormalities were assessed.
Time Frame: From the start of study drug administration upto Week 64
Population: As-treated population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants
  Atrial fibrillation | 1 | 0 | 2 | 0
  Atrial flutter | 0 | 1 | 0 | 0
  Bundle branch block left | 0 | 0 | 1 | 0
  Supraventricular extrasystoles | 1 | 0 | 0 | 0
  Tachycardia | 1 | 1 | 1 | 2

21. Secondary Outcome: Mean Serum Concentrations of MEDI9929
Description: The mean serum concentrations of MEDI9929 was observed at specified timepoints.
Time Frame: Week 0 (Day 1) to Week 64
Population: Pharmacokinetic population included all participants who received MEDI9929 and have a sufficient number of serum concentration measurements. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 133 | 128 | 132
ng/mL
  Week 4: number analyzed (Participants) | 129 | 126 | 130
  Week 4 | 3933.6 (3022.7) | 10733.1 (4649.4) | 39722.7 (15140.7)
  Week 12: number analyzed (Participants) | 129 | 121 | 126
  Week 12 | 6215.8 (3779.2) | 16625.4 (7751.6) | 63223.7 (60627.6)
  Week 20: number analyzed (Participants) | 126 | 113 | 116
  Week 20 | 6028.3 (2897.9) | 18237.1 (8721.9) | 64442.9 (22558.3)
  Week 28: number analyzed (Participants) | 127 | 117 | 120
  Week 28 | 6084.1 (2885.5) | 19373.4 (9191.4) | 64659.9 (24121.6)
  Week 40: number analyzed (Participants) | 127 | 117 | 118
  Week 40 | 6050.4 (3296.4) | 18926.1 (10252.7) | 64404.0 (26473.0)
  Week 52: number analyzed (Participants) | 128 | 118 | 116
  Week 52 | 6027.2 (3024.8) | 18821.9 (10435.2) | 68899.1 (71137.2)
  Week 64: number analyzed (Participants) | 123 | 116 | 113
  Week 64 | 632.8 (519.5) | 1991.2 (1882.4) | 6986.0 (5289.0)

22. Secondary Outcome: Number of Participants With Positive Antibodies to MEDI9929
Description: Blood samples for immunogenicity assessment included the determination of anti-drug antibodies (ADA) for MEDI9929. The number of participants with positive serum antibodies to MEDI9929 were presented.
Time Frame: Week 0 (Day 1) to Week 64
Population: As-treated population included all participants who received any study drug. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
Number analyzed (Participants) | 138 | 138 | 137 | 137
Participants
  ADA Positive at Baseline: number analyzed (Participants) | 138 | 137 | 136 | 135
  ADA Positive at Baseline | 7 | 1 | 2 | 2
  ADA prevalence: number analyzed (Participants) | 138 | 136 | 131 | 131
  ADA prevalence | 13 | 6 | 2 | 4
  ADA incidence: number analyzed (Participants) | 138 | 136 | 131 | 131
  ADA incidence | 13 | 5 | 1 | 3
  Neutralizing antibody- ADA Positive: number analyzed (Participants) | 138 | 136 | 131 | 131
  Neutralizing antibody- ADA Positive | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 upto Week 64
Arm/Group | Placebo | MEDI9929 70 mg | MEDI9929 210 mg | MEDI9929 280 mg
All-Cause Mortality (participants affected / at risk) | 0/138 | 1/138 | 0/137 | 0/137
Serious Adverse Events (participants affected / at risk) | 18/138 | 17/138 | 13/137 | 18/137
Other Adverse Events (participants affected / at risk) | 56/138 | 49/138 | 44/137 | 50/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=138) | MEDI9929 70 mg (N=138) | MEDI9929 210 mg (N=137) | MEDI9929 280 mg (N=137)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical leukoplakia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (23) | 5 (5) | 4 (4) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=138) | MEDI9929 70 mg (N=138) | MEDI9929 210 mg (N=137) | MEDI9929 280 mg (N=137)
Nasopharyngitis (Infections and infestations) | 16 (26) | 19 (24) | 19 (25) | 15 (30)
Headache (Nervous system disorders) | 6 (11) | 6 (10) | 11 (21) | 5 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 47 (111) | 31 (50) | 23 (37) | 35 (47)
Bronchitis (Infections and infestations) | 7 (11) | 7 (7) | 5 (6) | 9 (11)

LIMITATIONS AND CAVEATS:
A non-pre-specified statistical analysis was performed and generated the Measure of Dispersion for Outcome Measures 4 and 6.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.